CLINICAL TRIAL: NCT05882188
Title: Is, in Infertile Women Undergoing a Basic Fertility Work-up, Tubal Flushing With Oil-based Contrast Medium During Hysterosalpingography (HSG) Cost-effective Compared to Tubal Flushing by Hysterosalpingo-foam Sonography (HyFoSy)?
Brief Title: The Cost-effectiveness of Hysterosalpingography Versus Hysterosalpingo-foam Sonography During Fertility Work-up
Acronym: FOil
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. Velja Mijatovic, Professor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83352.018.22
Record Dates: First submitted 2023-05-05; First posted 2023-05-31 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Infertility
Keywords: Hysterosalpingography; Hysterosalpingo Foam Sonography; Infertility work-up; Cost-effectiveness; Live birth; Randomized controlled trial
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubal flushing during HSG with oil-based contrast (Experimental): Tubal flushing during HSG HSG will be performed by a gynaecologist, fertility doctor or nurse according to local protocols. HSG will be performed in the follicular phase of the cycle. Preferably, HSG is performed in the next cycle after randomization, but if this is not feasible the procedure may be postponed up till one month after randomization. After cleaning the vagina and cervix, a vacuum cervix adapter will be applied to the cervix or a Lipiodol resistant balloon catheter or hysterophore will be placed through the cervix. Up to 15ml of Lipiodol Ultra Fluid will be injected into the uterine cavity and its spread directly monitored by fluoroscopy. Six to eight radiographs will be taken and assessed by a gynaecologist or radiologist. The maximum amount of oil-based contrast medium is set at 15ml.
  Interventions: Procedure: Oil-based contrast
- Tubal flushing HyFoSy (Active Comparator): Tubal flushing during HyFoSy will be performed by a gynaecologist, fertility doctor, sonographer or nurse according to local protocols. HyFoSy will be performed in the follicular phase of the cycle. Preferably, HyFosy is performed in the next cycle after randomization, but if this is not feasible the procedure may be postponed up till one month after randomization. During HyFoSy approximately 5-10cc of foam will be introduced through a little cervical balloon-less applicator into the uterine cavity. During infusion of the foam into the uterine cavity, a transvaginal ultrasound will be performed which shows whether the Fallopian tubes are patent. The assessment of the procedure will be done by the one who performed the procedure.
  Interventions: Procedure: ExEm Foam

INTERVENTIONS:
Procedure: Oil-based contrast — oil-based contrast fluid, Lipiodol Ultra Fluid. Lipiodol is a solution of iodinated ethyl esters of fatty acids of poppyseed oil. Equivalent to 480 mg iodine per ml. The maximum dosage is 15ml. Lipiodol is produced by Guerbet, France. Lipiodol is FDA approved and registered as contrast agent for HSG.
  Arms: Tubal flushing during HSG with oil-based contrast
Procedure: ExEm Foam — ExEm Foam which is created by mixing 5ml ExEm-gel and 5ml of purified water. ExEm-gel contains hydroxyethylcellulose and glycerol. The ExEm Foam is distributed by IQ Medical Ventures, the Netherlands. ExEm Foam is FDA approved, CE marked and registered as contrast agent for HyFoSy.
  Arms: Tubal flushing HyFoSy

SUMMARY:
Hysterosalpingography (HSG) and hysterosalpingo-foam sonography are two methods to assess tubal patency during fertility work-up. This study aims to investigate the effectiveness of tubal flushing with oil-based contrast during HSG compared to tubal flushing during HyFoSy in women undergoing fertility work-up. The hypothesis is that tubal flushing with oil-based contrast during HSG leads to more live births than tubal flushing during HyFoSy.

DETAILED DESCRIPTION:
Background: The diagnostic work-up for infertility generally includes estimating the risk for tubal pathology and if indicated assessing tubal patency. Traditionally, tubal patency testing during the fertility work-up is performed with hysterosalpingography (HSG). In previous studies it has been demonstrated that tubal flushing with oil-based contrast during HSG resulted in more ongoing pregnancies than when HSG is performed with water-based contrast. HyFoSy is a more patient friendly alternative for HSG. Up till now, the fertility enhancing effect of tubal flushing with ExEm Foam during HyFoSy has only been studied in relatively small and observational studies.

Objectives:The main objective of this study is to determine whether tubal flushing with oil-based contrast during HSG results into more pregnancies leading to live births when compared to tubal flushing with ExEm Foam during HyFoSy, and whether this approach is cost-effective. In this study the safety of both strategies will also be compared.

Rationale: The hypothesis is that tubal flushing with oil-based contrast during HSG leads to more live births compared to tubal flushing with ExEm Foam during HyFoSy in women with an indication for tubal patency testing. If more live births are achieved, expensive fertility treatments will be less needed, which makes tubal flushing with oil-based contrast during HSG a cost-effective strategy.

Study design: This study is a multicenter randomized controlled trial with an economic analysis alongside it. Women with indication for tubal patency testing will be randomized to tubal flushing with oil-based contrast during HSG and tubal flushing with ExEm Foam during HyFoSy.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women or women with oligo-or anovulation
* Indication for tubal patency testing during the fertility work-up
* Sufficient understanding of the Dutch or English language
* Signed informed consent

Exclusion Criteria:

* Severe male factor with a total motile sperm count <3x106ml (pre-washed)
* Known contrast (iodine) allergy
* Women who have had a gynecologic procedure within the last 30 days
* Women with known or suspected reproductive tract neoplasia

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1102 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of pregnancies leading to live birth. | within six months after randomization
  Pregnancy is defined as a positive pregnancy test, increase in human chorionic gonadotropin (HCG) level or a pregnancy shown on ultrasonographic examination. Live birth is defined as the birth of live baby born beyond 24 weeks of pregnancy.

SECONDARY OUTCOMES:
Time to pregnancy leading to live birth | within six months after randomization
  Calculated from the day of randomization till the first day of the last menstrual bleeding before a positive pregnancy test.
Number of clinical pregnancies | within six months after randomization
  Clinical pregnancy is defined as gestational sac with or without heartbeat visible on ultrasound.
Number of miscarriages | within six months after randomization
  Miscarriage is defined as presence of non-vitality on ultrasound or spontaneous loss off pregnancy
Number of multiple pregnancies | within six months after randomization
  Multiple pregnancy is defined as two or more vital intrauterine pregnancies at 12 weeks gestation.
Number of ectopic pregnancies | within six months after randomization
  Ectopic pregnancy is defined as no intrauterine gestational sac with: an ectopic gestational sac OR HCG concentration >1500 international units per liter (IU/L) with free fluid/ectopic mass on ultrasound or serum HCG >2000IU/L without free fluid/ectopic mass on ultrasound
Number of adverse events | within one months after tubal patency testing
  e.g. infection, intravasation, thyroid dysfunction
Procedural pain scores | Within 15 minutes after tubal patency testing
  measured by Visual Analogue Scale (VAS) on a scale from 0.0 to 10.0 centimeter immediately after tubal patency testing.
Number of fertility treatment cycles | within six months after randomization
  e.g. intra uterine insemination, in vitro fertilization, intracytoplasmatic sperm injection
Number of pregnancy complications | within six months after randomization
  e.g. pregnancy induced hypertension, fetal growth restriction, still birth.
Cost-effectiveness | within six months after randomization
  Comparing the costs (including costs for tubal patency testing and additional fertility treatments) and the effects (chance of live birth)

CONTACTS AND LOCATIONS:
Locations (1):
- AmsterdamUMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamphuis D, Huijser JPM, van Welie N, Verhoeve HR, Kuijper E, de Bruin JP, van Dongen AJCM, Gielen SCJP, de Krom G, Janse F, Koks CAM, Nap AW, Anema JR, Bosmans JE, Stoker J, van Wely M, Mol BWJ, Mijatovic V, Dreyer K. Tubal flushing with oil-based contrast during hysterosalpingography versus tubal flushing by hysterosalpingo-foam sonography in infertile women undergoing fertility work-up: study protocol of a randomised controlled trial (FOil study). BMJ Open. 2024 Nov 24;14(11):e091778. doi: 10.1136/bmjopen-2024-091778. PMID 39581724